CLINICAL TRIAL: NCT03763357
Title: Acute Effects of Leg Heating on Skeletal Muscle Blood Flow in Patients With Symptomatic Peripheral Artery Disease
Brief Title: Acute Effects of Leg Heating on Skeletal Muscle Blood Flow
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain CT contrast from provider
Sponsor: Indiana University (Other)
Collaborators: Roseguini, Bruno, PhD (Individual); Purdue University (Other)
Responsible Party: Principal Investigator, Raghu Motaganahalli, Associate Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1809400414
Record Dates: First submitted 2018-11-23; First posted 2018-12-04 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Diathermy

STUDY DESIGN:
Intervention Model Description: All of the subjects in this study will receive leg heat therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heat Therapy (Experimental): Subject will dress in water-circulating trousers that are connected to a Heat Therapy (HT) pump. Warm water (42-43 degrees C) will be perfused through the pants for 90 minutes.
  Interventions: Device: Heat Therapy (HT)

INTERVENTIONS:
Device: Heat Therapy (HT) — Water at 42-43 degrees C will be circulated through the water circulating trousers to obtain calf skin temperature 39 degrees C followed by PET/CT imaging of generator-based 62Cu-ETS.

SUMMARY:
The purpose of this study is to apply local heat to the legs, thighs and buttocks of patients with peripheral arterial disease and use PET/CT imaging with an injectable stable radiotracer to study direct measurement of blood flow in the legs pre and post heat treatment.

DETAILED DESCRIPTION:
Cilostazol is the only effective medication available to treat walking pain (intermittent claudication) and it has multiple side effects. Overall improvement in walking performance in patients who use cilostazol is small. Endovascular and surgical interventions are effective alternatives for patients who don't respond to medical therapy, however, these procedures are costly and only applicable to patients with certain lesions types and carry a high risk of restenosis.

Heat therapy (HT) is an emerging non-invasive approach that has been shown to enhance vascular function of the leg in old individuals. The objective of this study is to test the hypothesis that a single session of heat therapy will increase local muscle tissue blood flow in the calf of patients with PAD as assessed by PET/CT imaging of generator-based 62Cu-ETS.

Subjects who have met inclusion criteria will volunteer for a single experimental visit. Participants will wear the water circulating pants and asked to rest supine for 30 minutes inside the scanner. Water at 43 degrees C will be perfused through the pants for 90 minutes with the goal to increase skin temperature in the calf to 39 degrees C. IV injections of 62Cu-ETS and subsequent perfusion imaging will be performed at the end of the 30 minute baseline period, after 45 minutes of heat therapy and at the end of the intervention (90 minutes). Due to the short half life of 62Cu, radioactivity from the prior administrations will not interfere with acquisition of a subsequent PET scan at this timing interval.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a stable symptomatic claudication for >/= 6 months
* Ankle brachial index < 0.9

Exclusion Criteria:

* Uncontrolled diabetes
* Heart failure
* COPD
* Critical limb ischemia
* Prior amputation
* Exercise-limiting co-morbidity
* Recent (< 3 months) intra-inguinal revascularization or planned in study period
* Plans to change medical therapy during duration of study
* Active cancer
* Chronic kidney disease (eGFR < 30)
* HIV positive, active HBV or HCV disease
* Presence of an clinical condition that makes the patient not suitable to participate in the trial
* Peripheral neuropathy, numbness or paresthesia in the legs
* Morbid obesity BMI > 36 or unable to fit into water-circulating pants
* Open wounds or ulcers on the extremity
* Claustrophobia/unable to tolerate PET/CT scanning
* Women of child-bearing age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in calf blood flow | Blood flow measurements will be completed at baseline (0 minutes) and after 45 and 90 minutes of exposure to heat therapy or a control regimen
  Calf muscle perfusion rate (mL⋅min-1⋅g-1) will be obtained after administration of tracer 62Cu-ETS before, during and after exposure to heat therapy or a control intervention. Changes from in perfusion rate from baseline to 45 minutes and 90 minutes of heating or control will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Raghu L Motaanahalli, MD, Principal Investigator — Indiana University

IPD SHARING:
Plan to Share IPD: No